CLINICAL TRIAL: NCT07279740
Title: Methylphenidate Primed iTBS for Apathy in Neurocognitive Disorders
Brief Title: Combined Brain Stimulation and Methylphenidate Treatment for Apathy in Dementia
Acronym: PRIME
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Alzheimer Society of Canada (Other); Sunnybrook Research Institute (Other); Brain Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SUN-6831
Record Dates: First submitted 2025-11-25; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Alzheimer s Disease; Alzheimer Dementia (AD); Alzheimer Dementia; Alzheimer Disease; Apathy; Apathy in Dementia
Keywords: apathy; dementia; Alzheimer's disease; methylphenidate; rTMS; iTBS; repetitive transcranial magnetic stimulation; intermittent theta burst stimulation
MeSH Terms: conditions — Alzheimer Disease; Lethargy; Dementia | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methylphenidate + iTBS (Experimental): Participants are currently receiving methylphenidate and receive iTBS in this study.
  Interventions: Device: intermittent theta burst stimulation (iTBS); Drug: Methylphenidate (MPH)
- iTBS only (Experimental): iTBS only, no medication for apathy
  Interventions: Device: intermittent theta burst stimulation (iTBS)

INTERVENTIONS:
Device: intermittent theta burst stimulation (iTBS) — iTBS is a form of repetitive transcranial magnetic simulation (rTMS), a non-invasive form of brain stimulation.
Drug: Methylphenidate (MPH) — Participants will be on methylphenidate clinically prior to the trial
  Arms: Methylphenidate + iTBS

SUMMARY:
This study evaluates whether the combined treatment of methylphenidate and non-invasive brain stimulation, called intermittent theta burst stimulation, can effectively treat apathy in individuals with Alzheimer's disease or mixed AD/vascular dementia

ELIGIBILITY:
Inclusion Criteria:

* Alzheimer's disease or mixed Alzheimer's disease and vascular disease
* MMSE score 10-28 inclusive
* Clinically significant apathy
* Stable dose of psychotropic medication
* Care partner must spend at least 10hrs/week with the participant

Exclusion Criteria:

* Major Depressive Episode
* Clinically significant agitation, delusions, hallucinations
* Currently talking a dopaminergic agent other than methylphenidate
* Failure to clear the TMS adult safety scale (e.g. unapproved pacemakers, metallic implants, history of epilepsy)
* Central nervous system abnormalities (other than Alzheimer's disease) deemed clinically significant by study physician or seizures
* Any condition that in the opinion of the study physician, makes it medically unsafe for the patient to enroll in the trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in Neuropsychiatric Inventory-Apathy (NPI-A) score | 2 weeks
  Assesses apathy total (frequency x severity) using the NPI-A based on scores provided by the care-partner through an interview with the assessor. Scores range from 0-12 with a higher score representing worse apathy.

CONTACTS AND LOCATIONS:
Overall Officials: Krista Lanctot, PhD, Principal Investigator — Sunnybrook Research Institute
Locations (1):
- Sunnybrook Research Institute, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided